CLINICAL TRIAL: NCT04618055
Title: A Prospective, Open Label, Randomized, Double Arm, Multicenter Study to Evaluate the Performance of NiTiDent Tuah Porous NiTi Dental Implants in Single Tooth Gap in the Posterior Mandible
Brief Title: Clinical Evaluation of NiTiDent Tuah Porous NiTi Dental Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nitium Technology Sdn Bhd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTSB/MD/01-01-CIP-01 version 1
Record Dates: First submitted 2020-11-02; First posted 2020-11-05 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Partial-edentulism
Keywords: Dental Implant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NiTiDent Tuah Porous NiTi Dental Implants (Experimental)
  Interventions: Device: NiTiDent Tuah Porous NiTi Dental Implants
- Control Implant (Active Comparator)
  Interventions: Device: Control Dental Implant Systems

INTERVENTIONS:
Device: NiTiDent Tuah Porous NiTi Dental Implants — A newly developed NiTiDent Tuah porous NiTi cylindrical bone level dental implant measuring 4.5 mm in diameter and 10 mm in length and an abutment system of different heights and angulations produced by Nitium Technology Sdn Bhd.
  Arms: NiTiDent Tuah Porous NiTi Dental Implants
Device: Control Dental Implant Systems — A market approved bone level dental implant systems measuring 4.5 mm in diameter and 10 mm in length and an abutment system of different heights and angulations
  Arms: Control Implant

SUMMARY:
The purpose of this prospective, open-label, randomized, double arm multicenter study is to evaluate the safety and clinical performance of a newly developed NiTiDent Tuah porous NiTi dental implant (from Nitium Technology Sdn Bhd) in singletooth gap in the posterior mandible 1 year after implant placement and 8 months after implant loading. Second, To investigate the clinical outcome of the interventional dental implant (NiTiDent Tuah Porous NiTi dental implant) compared to control dental implant. The hypothesis is set to no difference in the clinical outcome for the two types of implants based on the outcomes of the primary and secondary endpoints.

DETAILED DESCRIPTION:
The primary endpoint is to assess implant survival rate over a 12-month period. A surviving implant is defined as an integrated implant in the patient's jaw bone at the time of assessment. Secondary endpoints include the assessment of implant stability, crestal bone levels, peri-implant soft tissue conditions, implant success, and patient satisfaction and related outcomes over several intervals within a 12-month period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex and at least 18 years of age.
2. Ability to understand and provide informed consent before starting the study.
3. Ability and willingness to comply with all study requirements to be evaluated for each study visit.
4. The patient, if of child-bearing potential, has a negative urine pregnancy test.
5. Adequate oral hygiene to allow for implant therapy consistent with standards of care.
6. Adequate bone volume to accommodate the planned endosseous dental implant placement of 4.5 mm in diameter and 10 mm in length.
7. Adequate interocclusal distance (crown height space) of at least 6 mm measured from the alveolar crest to the occlusal table.
8. Intact buccal table as verified by Cone Beam Computed Tomography (CBCT). If absent, patient should be excluded from enrollment in the study.
9. One tooth in the posterior mandible (first or second molar) planned to be restored with a dental implant as determined by the patient's dental provider.
10. The site to be treated is surrounded by two natural teeth (one anterior and one posterior to it).
11. Primary stability of implant consistent with standards of care is achieved at the time of implant placement. Minimum primary stability, insertion torque at the value stated in the implants's Instructions for Use (IFU) (this will be a criterion that is met at the time of surgery).
12. Patients must be physically able to tolerate conventional surgical and restorative procedures.
13. Presence of opposing dentition with a functional occlusion.

Exclusion Criteria:

1. Presurgical

   * Patient reports tobacco uses within the last five years. Tobacco use for this study is defined as a current smoking habit with moderate or heavy smoking (more than 10 cigarettes per day) or tobacco chewing use.
   * History of alcoholism or drug abuse within the past 5 years.
   * Severe wear with an etiology of bruxism or clenching habits.
   * Patients in need of bone grafting at the site of the intended implantation site.
   * Patients who have previously failed implants at the site intended for study implant placement.
   * Patients in need of other treatments or surgeries at a site adjacent to the intended implantation site.
   * Patients with active infection or severe inflammation in the areas intended for implant placement.
   * Patient has significant untreated periodontal disease, severe recession, caries, clinical or radiographic signs of infection within two adjacent tooth positions of implant area.
   * History of HIV infection, Hepatitis B or C.
   * Patients has history of systemic disease that precludes standard dental implant therapy or alters daily activities to a level consistent with ASA (American Society of Anesthesiologists) III classification (including cardiovascular, hepatic, renal, gastrointestinal, metabolic, neurologic, pulmonary, endocrine, autoimmune, or psychiatric disorders).
   * Presence of local inflammation or mucosal diseases such as lichen planus.
   * Patient has history of consistent with high risk for subacute bacterial endocarditis.
   * Current hematological disorder or warfarin (or similar) therapy.
   * Patient has history of disease that affects bone metabolism, congenital connective tissue disorders (e.g., osteogenesis imperfecta), or Paget's disease.
   * Patient is taking medications or having treatments known to have an effect on bone turnover, including thiazide diuretics, calcitonin, systemic steroids, bisphosphonates, vitamin D (>800 IU/day), estrogen or progesterone therapy.
   * History of steroid treatment of duration of 2 weeks or longer in the past 2 years.
   * Patient currently undergoing chemotherapy.
   * Patient has history of radiation treatment to the head or neck.
   * Physical or mental handicaps that would interfere with patient's ability to exercise good oral hygiene on a regular basis.
   * Use of any investigational drug or device within the 30-day period immediately prior to implant surgery.
   * Patient is pregnant and lactating.
2. Post Implant Surgery:

   * Lack of implant primary stability.
   * Inappropriate implant position for prosthetic requirements.
   * Major simultaneous augmentation procedures at surgery.
   * X-ray not showing the implant from first bone contact to apical tip.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Implant survival | 12-month
  A surviving implant is an integrated implant in the patient's jaw bone at the time of assessment.

SECONDARY OUTCOMES:
Assess Implant Stability (Resonance Frequency Values) | Day 0 (Baseline), week 18, week 36 and week 52
  The measurement of Implant stability quotient (ISQ) value that indicates the level of stability and osseointegration in dental implants at the time of implant placement (Day 0 - 1st visit) and at 18 weeks (3rd visit), 36 weeks (5th visit) and 52 weeks (6th visit) after implant placement.
Crestal Bone Levels Evaluation | Day 0 (Baseline), week 22, week 36 and week 52
  The mesial and distal bone levels will be measured at baseline (during implant placement, Day 0 - 1st visit), at 22 weeks (during placement of the crown - 4th visit), 36 weeks (5th visit) and 52 weeks (6th visit) post implant placement by means of a single reader on standardized periapical radiographs.
Peri-Implant Soft Tissues Evaluation | Week 22, week 36 and week 52
  The conditions of the peri-implant soft tissues will be evaluated by probing depth, bleeding on probing, suppuration and dehiscence at 22-week (4th visit), 36-week (5th visit) and 52-week (6th visit) follow-up visit.
Implant Success Evaluation | 12-month
  Evaluation of implant success as assessed in the absence of post-surgery complications and other adverse events.

OTHER OUTCOMES:
Patient Satisfaction | Week 52
  Patient satisfaction will be assessed after 12 months of implant placement using a validated Patient Satisfaction Questionnaire (PSQ). The score on each question is divided into 6 scales with the lowest indicates "Extremely poor" while the highest indicates "Excellent".
Patient Related Outcome | Day 0 (Baseline) and week 52
  Patient related outcome will be assessed before and after 12 months using a validated OHIP-M. The data will be analysed including descriptive statistics (Chi-square test) for total patient sample and according to the two treatments groups (control and NiTi). Within the same group, mean and standard deviation for OHIP-14 scores (before and after the treatment) will be analysed using paired t-test, while independent t-test will be used to compare between the control and NiTi groups. The score on each question is divided into 5 scales with the lowest (1) indicates "Strongly agree" while highest (5) indicates "Strongly disagree".

CONTACTS AND LOCATIONS:
Overall Officials: Lim Tong Wah, BDS, Principal Investigator — Universiti Teknologi Mara
Locations (3):
- Malaysia (3):
  - Faculty of Dentistry, Universiti Kebangsaan Malaysia, Kuala Lumpur, Kuala Lumpur
  - Faculty of Dentistry, Universiti Malaya, Kuala Lumpur, Kuala Lumpur
  - Faculty of Dentistry, Universiti Teknologi MARA, Sungai Buloh, Selangor